Wayne Zhou, Ph. D.

Study: The Effects of OMT on the Expression of Immune Cell Biomarkers
Study Protocol

**Document Date: October 31, 2018** 

NCT03250312

# The Effects of Osteopathic Manipulation on the expression patterns of immune cell biomarkers

# 1. Specific Aims:

This proposal intends to study the effects of osteopathic manipulative treatment (OMT) on the biomarker expression patterns in human immune cells, by using the novel protein subcellular localization (PSL) microarray technology developed in Dr. Wayne Zhou's (PI) lab. The PSL microarray is the third generation of biochips (after DNA microarray, protein microarray) that can determine both the expression and subcellular localization protein profiling in high throughput screening format allowing for rapid identification of thousands of proteins. For the current study, we propose to use the PSL technology to determine the expression patterns of 60-400 cell surface proteins/biomarkers in human peripheral blood mononuclear cells (PBMC) of study participants with a history of low back pain, before and after OMT. We propose to identify and validate those proteins whose expression levels have been changed in most participants after OMT. From this study, we shall develop a platform to study the effects of different kinds of OMT techniques on participants with various types of pain conditions, and uncover the important immune cells that are affected by OMT techniques, therefore to uncover the molecular mechanisms of OMT.

Here are the specific aims for the current proposal:

Specific Aim 1: Determine the expression patterns of 60 surface biomarkers for human immune cells in PBMC of the participants, before and after OMT.

Specific Aim 2: Identify those specific proteins whose expression patterns have changed the greatest number of participants after OMT.

# 2. Research Strategy

**2-1. Significance:** Within the osteopathic profession most research on the effect of OMT on the immune system has involved lymphatic pump techniques. These techniques involve rhythmic compressions applied to the chest or abdomen, or through the lower extremities to maximize pressure gradients between the thorax and abdomen (page 632, 1). Studies performed in the 1920's and 30's found increases in serum leukocytes (2-3) and antibody titers (4) with splenic lymphatic pump techniques. Contemporary studies have detected changes in serum immune cell concentrations and inflammatory markers in response to lymphatic pump techniques. Mesina et al (5) measured blood cell counts following pectoral traction and splenic pump techniques and found significantly increased basophil counts in the 15-60 minute period post-treatment. However, there was individual variability with one subject demonstrating a significant increase persisting 4 hours post-treatment. Noll et al (6) found a decrease in serum platelet counts after participating nursing home residents received a single 6 minute OMT treatment consisting of lymphatic and myofascial techniques. Walkowski et al (7) found increases in serum cytokines, including IL-6, with a single 7-minute lymphatic treatment consisting of thoracic, splenic, and hepatic pump techniques. Licciardone et al (8) found several cytokines that were significantly associated with low back pain. Of these inflammatory markers, tumor necrosis factor concentrations significantly decreased after 12 weeks with 6 OMT sessions. These changes in serum immunologic factors

may be due to the OMT techniques' effect on the central lymphatic system. Lymphatic pump techniques have been shown to transiently increase central lymphatic flow, lymph leukocyte concentrations, and IL-6 concentrations (9-13).

Changes in lymphatic markers have been seen with other types of manual techniques. Soft tissue massage has been shown to significantly increase thymic and splenic T cell number in mice (14), increase serum natural killer cell and lymphocyte numbers in women with early stage breast cancer (15), and increase natural killer cell cytotoxicity in stable preterm infants (16). Serum from participants receiving spinal manipulation (HVLA) has been shown to significantly increase *in-vitro* immunoglobulin G and IL-2 synthesis in peripheral blood mononuclear cells (17-18). Spinal manipulation has also been shown to modify serum IL-6 levels (19) and decrease lymphocyte activation (20). The proposed study will expand upon the biomarker evidence base by investigating the effects of OMT on the biomarker expression patterns in serum immune cells using the PSL (protein subcellular localization) microarray technology.

The PSL (protein subcellular localization) microarray technology is the novel technology developed in Dr. Zhou's lab. It provides a unique approach to simultaneously determine subcellular localization and expression profiles of potentially thousands of proteins from one experiment. The technology has been already been used to identify the differences in protein expression between normal and cancer breast cell lines (21-23). The technology has also identified proteins with unique subcellular localization patterns between normal and cancer cells with breast origin and prostate origin (21-23).

**2-2. Innovation:** We propose to study the effects of OMT on serum immune cells using a system biology approach through the use of novel PSL microarray technology. No studies have yet investigated the effects of OMT using this technology, which may be able to detect changes in biomarker expression on immune cells even in the absence of cell concentration changes. We propose to use 40 participants for the experiments, 20 in the OMT group, and 20 in the control group. This number of participants should give us adequate statistical power to detect the difference in biomarker expression change. In addition, this proposal could provide a platform for future studies investigating the effects of different OMT techniques, and therefore to understand the molecular mechanism for OMT.

# 2-3. Preliminary data:

**2-3a.** Summary of the PSL microarray technology and its application on biomarker identification (Ref). The PSL microarray technology, also known as DAMA staining technology, is a novel technology that has combined the power of immunohistochemical staining and the parallel analysis of antibody microarrays (2123). It is equivalent to carry out 1000 immunostaining experiments from single immunostaining experiment. To our knowledge, this is the unique technology that can determine both the subcellular localization and expression profiles of thousands of proteins in high-throughput format.

Instead of capturing ligands on the array support like DNA microarray, PSL microarrays deliver multiple antibodies to their antigens in a position-addressable manner (Fig. 1). In this method, cells grown to the desired states on the cover slip, are fixed and permeabilized with standard methods (step 1). An array of antibodies on a membrane is then placed on the top of the cell with the antibodies facing the cells and incubated for an hour. During the incubation, antibodies dissociate from the array membrane and bind to their respective antigens in the cells without significant lateral diffusion (step 2). Afterward, the array membrane is removed, leaving the bound antibodies attached to the cellular antigens *in situ* (step 3). Enzyme-labeled secondary antibodies are then used to detect the bound primary antibodies on the cells (step 4). This way, the expression levels of multiple antigens can be determined simultaneously.

When fluorophore-conjugated secondary antibodies, instead of enzyme-labeled secondary antibodies, are used to detect the bound antibodies (step 4, Fig. 1), both the expression level and cellular localizations of multiple antigens can be determined using the fluorescent or confocal microscopes.



Fig. 1. Schematic representation of the PSL microarray technology

Identification of potential biomarkers for breast cancer by using the PSL microarray technology. (21) Dr. Zhou's lab has developed the PSL microarray technique and demonstrated its application on identifying the differentially expressed proteins between normal and cancer breast cell lines (4). For this purpose, protein expression profiles of ten different cell lines from human mammary glands were obtained using the PSL microarray technology and subjected to intensity integration and data analysis. Ten proteins were identified by DAMAPEP, (DAMA protein expression profiling, a software developed at his lab to retrieve, normalize, scale and analyze the intensity data), to have differential expression levels in cancer cells versus normal cells. Five proteins, RAIDD, Rb p107, Rb p130, SRF and Tyk2, were identified to have higher expression levels in cancer cells, and were confirmed by western blotting analysis (21).

Identification of potential biomarkers with different subcellular localizations for breast cancer and prostate cancer, by using PSL microarray technology (22-23). Dr. Zhou's lab has developed the PSL microarray technology that provides a new approach to the global analysis of protein subcellular localization (SCL) profiling in fixed cells. His lab has developed and optimized this technology, generated ChipView, a program for management and analysis of molecular image database, and utilized the technique to identify

proteins with unique SCL in breast cancer cell lines. The subcellular profile images of 360 proteins in a normal breast cells are shown in Fig 2a, and the subcellular localization profiles of the 360 proteins in two benign and seven carcinoma cells are shown in Fig 2b. From data analysis, a protein, Cyclin B1, was identified and validated with different SCLs between normal and cancer cell lines (22). Similar research has been carried out in prostate cancer and normal cell lines (23).



Fig 2. (A, left) Summary of representative molecular images of 360 proteins in one normal breast cell, as determined by the DAMA staining technology (22).

Each image represents the image of the corresponding protein in the tested sample. Images shown were taken with 63x objective lens. (B, right) Subcellular localization (SCL) profiles of 360 proteins in two benign and seven carcinoma derived cells, presented with a custom-defined color code scheme. Red indicates a protein is localized to the nuclei, green indicates a protein is localized to the cytoplasm, yellow indicates a protein is localized both to nuclei and in cytoplasm, and black represents an uncertain SCL for the protein.

Each column represents the SCL codes of the proteins in the same cell line, and each row represents the SCL codes of the same protein in different cell line samples.

2-3b. Summary of the funded study on "identify novel biomarkers for sDILI (severe Drug Induced Liver Injury) by using novel PSL microarray technology (was called DAMA staining technology). This grant proposal was funded by the Warner / Fermaturo research grant. Dr. Zhou's lab has studied the effects of different compounds on the expression profiles of 23 different Cytochrome P450s in HepG2 cells.

His lab has obtained 9 different compounds, 3 sDILI compounds (Ketoconazole, Troglitazone, Flutamide) and 6 non-sDILI compounds (Erythromycin freebase, Erythromycin estolate, SDS, Budesonide, Nicardipine, Olmesartan). The expression profiles of 23 different cytochrome P450s (CYPs) in the HepG2 cells treated with those compounds and controls are obtained and summarized in Fig 3. Unfortunately, no differentially expression changes for any P450 subtype proteins were observed between cells treated with different concentration (40 M and 80 M) of sDILI compounds and non-sDILI compounds.

Treatment of flutamide has been reported to increase the expression of liver cytochrome P450 1A2 (24). Therefore, his lab has determined the expression profiles of 23 different cytochrome P450s in the HepG2 cells treated with different concentration of Flutamide, (0 - 250 M) (Fig 4). No increase of cytochrome P451A2 was observed either.



Fig. 3. The expression profiles of 23 CYPs in HepG2 cells treated with different compounds and control (#0). The expression profiles were determined in triplets.



Fig. 4. The expression profiles of 23 CYPs in HepG2 cells treated with different concentration of Flutamide. The expression profiles were determined in triplets, and each experiment was repeated at least twice.

# 2-4. Approach:

# Specific Aim 1. Determine the expression pattern of 60 surface biomarkers for human immune cells in PBMC of participants, before and after OMT.

Experimental design: This prospective, randomized, controlled trial is proposed to investigate the expression patterns of  $\sim 60$  cell surface proteins in human immune cells, in the peripheral blood mononuclear cells (PBMC) of each participant, before and after intervention – OMT or seated control. This study will utilize participants with a history of low back pain (LBP) because several studies have demonstrated that patients with LBP have a significantly greater incidence and severity of somatic dysfunction than people without LBP (12, 26-27). Somatic dysfunction is the clinical indication of OMT, therefore participants with more somatic dysfunction may have a greater response to OMT than participants with less somatic dysfunction.

The study will be conducted over the course of one year. Forty men and women ages 20 to 65 years with at least one or more episodes of LBP in the past two weeks will be randomly assigned into one of two groups – control or OMT groups. Twenty participants will be assigned to each group. The study will begin recruitment in July 2017 pending institutional review board approval. Participants will be recruited from the surrounding Kirksville

area. Individuals who cannot tolerate OMT or have coagulation disorders will be excluded. Potential participants will be excluded from the study if they have had nonsteroidal antiinflammatory medication in the 48 hours prior to the study or if they have had corticosteroids in the 2 weeks prior to the study. Participants will be randomly assigned into two groups, control or OMT using a random number generator. Males and females will be randomized separately to ensure equal distribution into the two study groups. Demographics including sex, age, and body mass index (BMI) will be collected on all participants. All participants will receive two blood draws: first blood draw prior immediately prior to intervention and second blood draw following the intervention.

**OMT intervention:** The OMT treatment will begin with a brief physical examination to identify somatic dysfunction that the treating physician judges to be relevant to the individual participant's low back pain. OMT will be performed to improve the somatic dysfunctions that the treating physicians finds most relevant. The types of OMT techniques used will include muscle energy, articular, or high velocity-low amplitude (HVLA) as indicated by the physical findings and will be at the discretion of the treating physician. Additional techniques such as still, counter strain, facilitated positional release, balanced ligamentous tension, and cranial techniques may also be used at the discretion of the treating physician. The treatment will conclude with 2 minutes of pedal lymphatic pumping technique. The total treatment time will not to exceed 20 minutes. To encourage participation in the proposed study, participants who are assigned to the control group will have an opportunity to receive OMT after the second blood draw.

Control protocol: The control group will wait in another room for approximately 30 minutes.

**PBMC cell isolation.** PBMC cells will be isolated and prepared according to the company protocol which is summarized as below. Venous blood will be collected via venipuncture into the Vacutainer CPT tube (BD Biosciences). CPT tubes will be centrifuged at  $1800 \times g$  for 20 minutes at room temperature. After centrifugation, CPT tubes will be brought to a biological safety cabinet and carefully opened. The PBMC cells, which are in the layer just under the plasma (Figure 5), will be transferred to a 15 ml conical tube. The conical tubes will be centrifuged at  $250 \times g$  for seven minutes at room temperature. The PBMC cells will be re-suspend at  $5 \times 10^6$  viable lymphocytes per ml in PBS buffer.



Fig 5. Typical PBMC layers after centrifugation in BD Vacutainer CPT tube Fig 6 Diagram for the PSL microarray. Different color corresponds to different



lymphocytes, # corresponding to CD#

Coverslip preparation. 1004 of the suspended PBMC cells will be added to a poly-lysine coated coverslip (22 mm x 22 mm), and dried for 10-20 minutes at room temperature. The cells attached to the coverslips will be washed three times in PBS, and fixed with 4% paraformaldehyde in PBS. The detail protocol would be modified and optimized in the experiments.

Antibody selection and microarray preparation. The goal of this project is to purchase ~60 antibodies, which are the surface biomarkers for different human immune cells. We shall determine the expression patterns of the 60 proteins in the PBMC cells from the participants, before and after the OMT treatment by using the PSL microarray. The proteins with differentially expressed level after the OMT treatment will be identified from data mining and statistical analysis.

We plan to first purchase 30 antibodies, which are the biomarkers for different human lymphocytes. The selected antibodies and their major expression in different lymphocytes are summarized in Table 1. The PSL microarrays containing those antibodies will be made according the design in figure 6 by using the purchased antibodies and the nanoplotter at ATSU, and will be used for the proposed research. Most of the 30 proteins shown in Table 1 are expressed in 1-2 kinds of different lymphocyte cells. An increase or decrease in expression of those proteins could be related to the increase or decrease of the specific types of lymphocytes, which could provide potential mechanism for OMT on immune system activity.

The second set of 30 antibodies will be selected from the ~150 surface proteins summarized in the Appendix (with their expression patterns in human immune cells) and purchased later pending the findings from the analysis of the first 30 antibodies. The samples will be saved and stored in liquid nitrogen and retested for the second set of 30 antibodies.

The long-term plan. The long-term plan of the proposal is develop a research methodology for study the effect of OMT on immune system activity. The goal of the current proposal is to generate preliminary data, so that we could apply for the NIH grant to determine the expression patterns of 150-200 cell surface biomarkers for human immune cells in the PBMC cells of the participants, before and after OMT. For this purpose, a grant application based on the preliminary data generated from the current proposal will be submitted to NIH or AOA. Additional antibodies, as those listed in the Appendix, will be purchased if funded. The microarray containing 150-200 antibodies will be made similar to those used in the publication (23), and used for the longterm research.

Table 1. Summary of Antibodies used for the research and their expression in immune cells

| Markers | B Cells | Myeloid and mast | IK<br>ell | S | T Cells |
|---------|---------|------------------|-----------|---|---------|
|---------|---------|------------------|-----------|---|---------|

# Wayne Zhou, Ph. D.

| Cell Types | Antibody | Plasma<br>CEo<br>B Cells | <sub>S</sub> sir | nophil<br>Base | | ophil<br>Monocy | :e<br>IK<br>Vell | | <b>eleGtor y</b> nemory Cl<br>ell<br>T Cell | D8<br>T cell |
|---|---|---|---|---|---|---|---|---|---|---|
| Total B cell | BCR | Х | | | | | | | | |
| | CD19 | X | | | | | | | | |
| | CD20 | x | | | | | | | | |
| | CD138 | х | | | | | | | | |
| Eosinophil | CD9 | | Х | | | | | Х | | |
| | CD32 | X | X | | | Χ | | | | |
| | Siglec -8 | | Х | | Х | | | | | |
| Neutrophil | CD13 | | | Χ | | | | Х | | |
| | CD15 | | | Χ | | | | | | |
| | CD33 | | | Χ | Χ | Х | | | | |
| Basophil | CD123 | | | | X | X | | | | |
| Вазории | 1/2 - Ser | | | | Х | Λ | | | | |
| | Fc□ | | | | | | | | | |
| | R1 <sup>□</sup> | | | | Χ | | | | | |
| Monocyte | CD11b | Х | | | | Χ | Х | Х | | |
| | CD11c | Х | | | | Χ | Х | Х | | |
| | CD14 | Х | | | | Χ | | | | |
| | CD163 | X | | | | Х | | | | |
| NK cell | CD57 | | | | | | Х | | | |
| | CD335 | | | | | | Х | | | |
| | CD336 | | | | | | x | | | |

Program Director/Principal Investigator (Last, First, Middle): G. Wayne Zhou, Ph. D.

| | CD337 | | | Χ | | | | | | |
|--------|------------|---|---|---|---|---|---|---|---|---|
| T cell | CD3 | | | | Х | Х | Х | Х | Х | Х |
| | TCR 🗆 🗆 🗆 | | | | Х | | X | Χ | Χ | Х |
| | TCR 🗆 🗆 🗆 | | | | Х | Х | | | | |
| CD4 | CD4 | | Х | | | | Χ | Χ | | |
| | CD45RA | x | Х | | | | Χ | | | |
| | CR45RO | x | Х | | | | | X | | |
| CD8 | CD8 | | | X | | | | | Χ | Χ |
| | CD25 | | Χ | | | | | Χ | | |
| | Granzyme A | | Χ | | | | | | | Χ |

Determination of the expression profiles of the lymphocyte biomarkers in the PBMC cells. We propose to use similar approach as the published one (21) (also was summarized in the preliminary studies section B3) to determine the expression profiles of the 60 lymphocyte biomarkers in the PBMC cells, before and after the OMT. In summary, the PSL microarray containing the biomarkers will be put on top of the fixed PBMC cells, and incubated for 2 hours at the room temperature. The antibodies will be delivered to the targeted PBMC cells without diffusion. The sample will be washed three times in PBS (phosphate-buffered saline) to remove the unbound antibodies. The bound antibodies will be detected by alkaline phosphatase-conjugated secondary antibodies, followed with 1-step NBT/BCIP (nitro blue tetrazolium/5-bromo- 4-chloro-3-indolyl phosphate) substrate (Pierce). Images of protein expression profiles will be scanned by Brother MFC-7365DN scanner, and processed by Photoshop for intensity integration. The expression profile of 23 Cytochrome P450 in HepG2 cells is as shown in Figure 8. The expression profile of the lymphocyte biomarkers in the PBMC samples of the participates would be similar to those







Figure 9. The bound antibodies (Actin, row 1/3; GADPH row Figure 8. The expression profile of 23 CYPs in HepG2 cells are shown in 2/4) detected by with DyLight 680 (right) and DyLight 800 (left) triplicate. antibodies

(Fig 8)

The biomarker expression profiles in the PBMC cells can also be detected by the fluorescence-conjugated secondary antibodies. A protocol has been developed to detect the bound antibodies at 680nm and 800nm, by using the DyLight-680 conjugated secondary antibody and the DyLight-800 conjugated antibody (Rockland Antibody), respectively (Figure 9). The images show the bound antibodies for Actin (row 1 and 3), and for GADPH (row 2 and 4) on HTB129 cells, a breast cancer cell, obtained by Odyssey Imaging Systems. Both methods will be used to analyze biomarker expression patterns in the proposed study to identify the more effective method for future experiments.

<u>28</u>

OMB No. 0925-0001/0002 (Rev. 03/16 Approved Through 10/31/2018) Page \_\_\_ Continuation Format Page Specific Aim 2. Identify those specific proteins whose expression patterns have changed in the greatest number of participants after OMT.

**Sample Size.** To estimate the sample size needed to detect a mean difference of 0.5 in ratio of intensity (After/Before) between the OMT and in the control group, standard deviations of intensity (After/Before) in the two groups were estimated using PSL microarray staining, by using the data similar to the images shown in Figure 4. The data integration was carried out for each image by using the ScanAlyze in Image J, the intensity integration programs for DNA and protein microarray analysis. As summarized in Table 2, the mean ratio in the Control group is 1.32 with standard deviation of 0.34 and mean ratio in the Intervention group is 1.42 with standard deviation of 0.32 (28). Those data have been used to calculate the sample size needed for the proposed study as described below.

Table 2 Summary data from PSL Microarray Analysis

| Group | # Obs Mean | | Std Dev | Median |
|--------------|------------|------|---------|--------|
| Control 4 | | 1.32 | 0.34 | 1.20 |
| Intervention | 6 | 1.42 | 0.32 | 1.43 |

**Group sample size calculation.** Sample size calculations based on the data summarized in Table 2 reveal that recruiting a total 22 participants, 11 in the OMT group and 11 in the control group, will allow us to detect a difference of 0.5 in intensity (After/Before) in the two groups with a power of 0.92 at a significance level of 0.05, using two sample *t*-tests with unequal variances. We propose to use 40 patients for the experiments, 20 in the OMT group, and 20 in the control group. Therefore, we should have an adequately powered study.

**Data Extraction and data analysis.** The expression profiles of 60 biomarkers in the PBMC samples obtained by the PSL microarray staining, will be extracted by the program ScanAlyze of ImageJ, from the images similar to the above figures. The ratio change of every biomarker protein in PBMC samples, before and after the OMT will be analyzed by DAMAPEP, a software developed at the PI's lab to retrieve, normalize, and scale the data from

the exported intensity integration files. The mean change in intensity (After/Before) of biomarker expression for each of the 60 biomarkers will be compared between the OMT and control group using two sample *t*-test and biomarkers whose expression has changed significantly between the two groups will be identified. If needed, modification on published data analysis protocol and software in the paper (21) will be carried out for the project in order to identify the proteins with statistically meaningful expression change between the OMT group and the control group. The comparison would eliminate and normalize the expression change of biomarkers due to fluctuation and personal variation, and identify those differentially changed biomarkers due to the OMT.

**Potential Limitations**: The purposed study is investigating the impact of OMT on immune cell biomarkers. OMT can be accomplished with a wide variety of techniques. Most studies investigating the effect of OMT on immune cells use lymphatic pump OMT techniques. Other types of OMT techniques may not have the same effect. The purposed study will use a wide variety of OMT techniques consistent with what a patient with low back pain would receive in a clinical setting and conclude the treatment with a lymphatic pump OMT technique. Therefore, the current design will not allow for conclusions about the effect of any specific type of technique. Future studies will investigate the effect of different types of OMT techniques on the immune cell biomarkers.

Another potential limitation is that the method could be not sensitive enough to detect changes in biomarkers after 30 minutes post OMT. If no changes are seen during the initial investigation we will modify the protocol to increase the sensitivity of the technology or try different OMT techniques.

# 3. Bibliography and References

- 1. Kuchera ML. Lymphatics approach. In: Chila AG, ed. Foundations of Osteopathic Medicine. 3rd ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2011:786-808.
- 2. Castlio Y, Ferris-Swift L. Effects of splenic stimulation in normal individuals on the active and differential blood cell counts and the opsonotic index. Kansas City Coll Osteopath Surg 1932;16:10–6
- 3. Castlio Y, Ferris-Swift L. The effect of direct splenic stimulation on the cells and antibody content of the bloodstream in acute infectious disease. Kansas City Coll Osteopath Surg 1934;18:196–211
- 4. Lane MA. On increasing the antibody content of the serum by manipulation of the spleen. J of Osteopath 1920;27:361–4
- 5. Mesina J, Hampton D, Evans R, Ziegler T, Mikeska C, Thomas K, Ferretti J. Transient basophilia following the application of lymphatic pump techniques: a pilot study. J Am Osteopath Assoc 1998;98:91–4
- 6. Dons'koi B, Chernyshov V, Osypchuk D, Baksheev S. Repeated cupping manipulation temporary decreases natural killer lymphocyte frequency, activity and cytotoxicity. Journal Of Integrative Medicine [serial online]. May 2016;14(3):197-202. Available from: MEDLINE Complete, Ipswich, MA. Accessed January 5, 2017.
- 7. Walkowski S, Singh M, Puertas J, Pate M, Goodrum K, Benencia F. Osteopathic manipulative therapy induces early plasma cytokine release and mobilization of a population of blood dendritic cells. PLoS One. 2014 Mar 10;9(3):e90132. doi: 10.1371/journal.pone.0090132. eCollection 2014.

- 8. Licciardone JC, Kearns CM. Somatic dysfunction and its association with chronic low back pain, backspecific functioning, and general health: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012;112(7):420-428.
- 9. Knott EM, Tune JD, Stoll ST, Downey HF. Increased lymphatic flow in the thoracic duct during manipulative intervention. J Am Osteopath Assoc 2005;105:447–56
- 10. Hodge LM, King HH, Williams AG Jr, Reder SJ, Belavadi TJ, Simecka JW, Stoll ST, Downey HF. Abdominal lymphatic pump treatment increases leukocyte count and flux in thoracic duct lymph. Lymphat Res Biol 2007;5:127–33
- 11. Hodge LM, Bearden MK, Schander A, et al. Lymphatic Pump Treatment Mobilizes Leukocytes from the Gut Associated Lymphoid Tissue into Lymph. Lymphatic Research and Biology. 2010;8(2):103-110. doi:10.1089/lrb.2009.0011.
- 12. Schander A, Downey H, Hodge L. Lymphatic pump manipulation mobilizes inflammatory mediators into lymphatic circulation. Experimental Biology And Medicine (Maywood, N.J.) [serial online]. January 2012;237(1):58-63. Available from: MEDLINE Complete, Ipswich, MA. Accessed December 5, 2016.
- 13. Schander A, Padro D, King HH, Downey HF, Hodge LM. Lymphatic Pump Treatment Repeatedly Enhances the Lymphatic and Immune Systems. Lymphatic Research and Biology. 2013;11(4):219-226. doi:10.1089/lrb.2012.0021.
- 14. Major B, Rattazzi L, Brod S, Pilipović I, Leposavić G, D'Acquisto F. Massage-like stroking boosts the immune system in mice. Scientific Reports [serial online]. June 5, 2015;5:10913. Available from: MEDLINE Complete, Ipswich, MA. Accessed January 5, 2017.
- 15. Hernandez-Reif M, Field T, Fraser M, et al. Natural killer cells and lymphocytes increase in women with breast cancer following massage therapy. The International Journal Of Neuroscience [serial online]. April 2005;115(4):495-510. Available from: MEDLINE Complete, Ipswich, MA. Accessed January 5, 2017.
- 16. Ang J, Lua J, Shankaran S, et al. A randomized placebo-controlled trial of massage therapy on the immune system of preterm infants. Pediatrics [serial online]. December 2012;130(6):e1549-e1558. Available from: MEDLINE Complete, Ipswich, MA. Accessed January 5, 2017.
- 17. Teodorczyk-Injeyan J, Injeyan H, McGregor M, Harris G, Ruegg R. Enhancement of in vitro interleukin2 production in normal subjects following a single spinal manipulative treatment. Chiropractic & Osteopathy [serial online]. January 2008;16:1. Available from: Publisher Provided Full Text Searching File, Ipswich, MA. Accessed January 5, 2017.
- 18. Teodorczyk-Injeyan J, McGregor M, Ruegg R, Injeyan H. Interleukin 2-regulated in vitro antibody production following a single spinal manipulative treatment in normal subjects. Chiropractic & Osteopathy [serial online]. September 8, 2010;18:26. Available from: MEDLINE Complete, Ipswich, MA. Accessed January 5, 2017.
- 19. Roy R, Boucher J, Comtois A. Inflammatory response following a short-term course of chiropractic treatment in subjects with and without chronic low back pain. Journal Of Chiropractic Medicine [serial online]. September 2010;9(3):107-114. Available from: CINAHL Plus with Full Text, Ipswich, MA. Accessed January 5, 2017.
- 20. Davison S, Parkin-Smith G. The possible effect of upper cervical chiropractic manipulation on short-term lymphocytic response: a pilot study. European Journal Of Chiropractic [serial online]. October 2003;51(1):19-28. Available from: CINAHL Plus with Full Text, Ipswich, MA. Accessed January 5, 2017.
- 21. Song, X., Fu, G., Yang, X., Wang, J., Jiang, Z. and Zhou, G. W. (2008) "Protein expression profiling of breast cancer by DAMA (Dissociable Antibody Microarray) staining". *Mol Cell Proteomics*. 7, 163-169

- 22. Fu, G., Song, X., Yang, X., Peng, T., Wang, J., and Zhou, G. W. (2010) "Protein Subcellular localization profiling of breast cancer by using DAMA (Dissociable Antibody Microarray) staining". *Proteomics* 10, 1539-1544
- 23. Fu, G., Song, X., Yang, X., Mo, Y. and Zhou, G. W. (2016) "Protein subcellular localization profiling of prostate cell by DAMA (Dissociable Antibody Microarray) staining technology", *J. Proteomics & Bioinformatics*, 9: 001-008. doi:10.4172/jpb.1000382.
- 24. Wang, H. X, Liu, X., Xu, C. J., Ma, X. C, Long, J. E. and Li, D. (2005) "Induction of liver cytochrome P450 1A2 expression by flutamide in rats" *Acta Pharmacol Sin.* 11, 1382-6.
- 25. Gerets, H., H. J., Tilmant, K., Gerin, B., Chanteux, H., Depelchin, B. D., Dhalluin, S. and Atienzar, F. A. (2012) "Characterization of primary human hepatocytes, HepG2 cells, and HepaRG cells at the mRNA level and CYP activity in response to inducers and their predictivity for the detection of human hepatotoxins" *Cell Biol Toxicol.* **28:** 69–87.
- 26. Snider KT, Johnson JC, Degenhardt BF, Snider EJ, Burton DC. Association of low back pain, somatic dysfunction, and lumbar bone mineral density: reproducibility of findings. J Am Osteopath Assoc. 2014;114(5):356-367.
- 27. Snider KT, Johnson JC, Snider EJ, Degenhardt BF. Increased incidence and severity of somatic dysfunction in subjects with chronic low back pain. J Am Osteopath Assoc. 2008;108(8):372-378.
- 28. Zar, Jerrold H. 1984. Biostatistical Analysis (Second Edition). Prentice-Hall. Englewood Cliffs, New Jersey
- 29. Julious, S. A. 2010. Sample Sizes for Clinical Trials. Chapman & Hall/CRC. Boca Raton, FL.
- 30. Chow, S.-C., Shao, J., and Wang, H. 2008. Sample Size Calculations in Clinical Research (Second Edition). Chapman & Hall/CRC. Boca Raton, FL.
- 31. Machin, D., Campbell, M., Fayers, P., and Pinol, A. 1997. Sample Size Tables for Clinical Studies, 2ndEdition. Blackwell Science. Malden, MA.

### 4. PROTECTION OF HUMAN SUBJECTS

#### 4.1 DETAILED DESCRIPTION OF THE PROPOSED INVOLVEMENT OF HUMAN SUBJECTS

The proposed study will involve 40 participants receiving two venous blood draws; one blood draw immediately before and one immediately after the intervention. Twenty participants will receive OMT for up to twenty minutes as part of the protocol with the remaining 20 participants receiving OMT if desired.

# 4.2 SOURCES OF RESEARCH MATERIAL

a. Demographic information and past medical history. Basic demographic information and past medical history including frequency of low back pain will be collected from participants.

b. Surface protein expression of 60 cell surface proteins in human immune cells, in the peripheral blood mononuclear cells (PBMC) of each participant will be analyzed from peripheral blood before and after intervention.

# 4.3 RECRUITMENT AND INFORMED CONSENT

Participants will be recruited from the surrounding Kirksville area. A research investigator or their assistant will review the study with a potential participant, determine the participant's eligibility, and obtain informed consent using an informed consent document that will be reviewed and approved by the Institutional Review Board for ATSU-Kirksville pending study funding. The study will be registered with ClinicalTrials.gov.

#### 4.4 POTENTIAL RISKS

#### 4.4.1 PHYSICAL RISKS

The physical risks to the participant include the OMT and venous blood draws. The participant may feel some post-treatment soreness from the OMT and they may experience bruising from the blood draws. 4.4.2 PSYCHOLOGICAL RISKS

There are no psychological risks to the participant from the OMT or blood draws.

#### 4.4.3 SOCIAL RISKS

There are no social risks to the participant from the OMT or blood draws. The health information obtained during the study will be kept in a locked file cabinet and information used in this study will be de-identified prior to data analysis and results dissemination.

# 4.4.4 ECONOMIC RISKS

There are no economic risks to the participant from the OMT or blood draws.

#### 4.4.5 LEGAL RISKS

There are no legal risks to the participant from the OMT or blood draws.

# 4.5 ALTERNATIVE PROCEDURES OR THERAPIES

The participant may choose not to participate in the study.

# 4.6 PROCEDURES FOR PROTECTING AGAINST RISKS

Any residual soreness that a participant experiences from the OMT or blood draws is likely to be insignificant, though the participant may contact the Dr Karen Snider for options regarding care. The results of this research may be published; however, neither participants' names nor identities will be revealed, and records will remain confidential. Confidentiality will be maintained by using coded identification numbers on all forms. All consent forms and study data will be kept and treated as personal medical records. Only the investigators and study personnel will have access to this information. As required by Federal law, all personal health information will be maintained in accordance with the Health Insurance and Portability and Accountability Act (HIPAA) to ensure privacy.

# 4.7 RISKS AND BENEFITS TO SUBJECTS

#### 4.7.1 POSSIBLE BENEFITS TO SUBJECT

There are minimal risks to the participants. The minimal risks to the participants are reasonable compared to the knowledge to be gained from the proposed study and the benefit to the osteopathic profession. The participants may benefit from the OMT with regards to their low back pain, though treatment for low back pain is not an intended outcome.

# 4.7.2 POSSIBLE BENEFITS TO SOCIETY

The benefit to society will be the information obtained regarding the possible effects of OMT on immune biomarker expression. This knowledge can be integrated into the training of future osteopathic physicians.

# 5. DATA SAFETY MONITORING PLAN

Not applicable.

# **6 INCLUSION OF WOMEN AND MINORITIES**

Women and minorities are encouraged to participate in the proposed study.

# 7. TARGETED/PLANNED ENROLLMENT TABLE

| Time | # patients |
|----------|------------|
| Q4, 2017 | 10 |
| Q2, 2018 | 30 |
| Total | 40 |

| Program Director/Principal Investigator (Last, First, Middle): <u>G. Wayne Zhou, Ph. D.</u> The first set of 10 participants samples will be saved and retested with the second set of 30 antibodies. |
|---|
| 8. INCLUSION OF CHILDREN |
| Children are excluded from this study. |
| 9. VERTEBRATE ANIMALS |
| Not applicable |
| 10. SELECT AGENT RESEARCH |
| Not applicable |
| 11. MULTIPLE PD/PI LEADERSHIP PLAN |
| Not applicable |
| 12. CONSORTIUM/CONTRACTUAL ARRANGEMENTS |
| Not applicable |

# 13. LETTERS OF SUPPORT (E.G., CONSULTANTS)

Not applicable

# 14. RESOURCE SHARING PLAN

The research findings from this study are expected to be published in JAOA. Travel funds for presentation of the study findings have been requested to attend OMED in 2018.

| | Program Director/Principal Investigator (Last, First, Middle): | G. Wayne Zhou, Ph. D. |
|---|---|---|
| <del></del> | 20 | |



To view our full range of antibodies visit bio-rad-antibodies.com/immunology

Bio-Rad Laboratories, Inc.



**Appendix**